CLINICAL TRIAL: NCT06264687
Title: Serum Hepcidin Response After Intravenous Iron Therapy
Brief Title: Hepcidin After Intravenous Iron Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Pierre-Alexandre Krayenbühl (Other)
Responsible Party: Sponsor-Investigator, Pierre-Alexandre Krayenbühl, Clinical Professor, Hausarztpraxis Brauereistrasse
Organization: Hausarztpraxis Brauereistrasse (Other)
Other Study IDs: HepcidinIVIron
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Iron Deficiency (Without Anemia)
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the hepcidin hormone response after intravenous iron administration.

DETAILED DESCRIPTION:
Intravenous iron is often administered when peroral iron is insufficient to correct iron-deficiency or not tolerated. Few studies have shown a relationship between pretherapeutic serum hepcidin levels and response to intravenous iron infusion: the lower the pre-infusion hepcidin level, the fewer red blood cell concentrates were used to correct anaemia. However, there are no studies investigating hepcidin levels after intravenous iron supplementation. Furthermore, some studies showed an increase in hepcidin 24 hours after ingesting oral iron supplements, impairing the iron uptake the next day. However, how long hepcidin is increased after intravenous iron administration is unknown. Prolonged serum hepcidin concentrations after an iron infusion would reduce intestinal iron absorption and continued, simultaneous oral iron therapy would be pointless.

This study investigates whether and how serum hepcidin concentrations change after intravenous iron therapy. Women with iron deficiency (serum ferritin below 30ng/ml) without anaemia (hemoglobin >117g/l) receive 500mg iron (Ferinject®) intravenously. Serum hepcidin levels are measured before therapy (day 0) 2 days (day 2) and 7 days (day 7) after infusion.

ELIGIBILITY:
Inclusion Criteria:

* informed consent as documented by signature
* iron-deficiency (serum ferritin <30ng/ml)
* female gender
* premenopausal
* age >18 years
* body mass index (BMI) in normal range (18-25 kg/m²)
* the participant is linguistically and cognitively able to understand the study procedure

Exclusion Criteria:

* anaemia (hemoglobin <117g/l)
* allergy or contraindications for iron infusions
* anamnestic current pregnancy
* breastfeeding
* chronic inflammatory diseases (e.g. colitis)
* liver disease (alanine transaminase (ALT) >35 U/l)
* increased C-reactive protein (CRP) (>5mg/l)
* intake of dietary supplements containing iron (last 7 days)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: iron deficient non-anemic women
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Serum Hepcidin Change | 1 week
  The change of serum hepcidin levels over time (days 0, 2, 7) after intravenous iron administration.